CLINICAL TRIAL: NCT04473651
Title: Interventional, Randomized, Double-blind, Placebo-controlled, Sequential-group, Single-ascending Oral Dose Study Investigating the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Properties of Lu AG06479 and Open-label Cross-over Study to Investigate Intra-subject Variability and Effect of Food in Healthy Young Men
Brief Title: Safety and Tolerability of Lu AG06479 in Healthy Young Men
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for strategic reasons.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18452A
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single dose of Lu AG06479 or Placebo (Experimental)
  Interventions: Drug: Lu AG06479; Drug: Placebos
- Part B: Repeated dose of Lu AG06479 and Food interaction (Experimental): Sequence B1: Fed - Fasting - Fasting
  Sequence B2: Fasting- Fed - Fasting
  Sequence B3: Fasting- Fasting - Fed
  Interventions: Drug: Lu AG06479

INTERVENTIONS:
Drug: Lu AG06479 — capsules, orally (Part A and B)
  Other Names: ABX-1762
Drug: Placebos — Placebo - capsules, orally (Part A only)
  Arms: Part A: Single dose of Lu AG06479 or Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of Lu AG06479 and what the body does to Lu AG06479 after swallowing single doses of the drug.

DETAILED DESCRIPTION:
Part A: randomized, sequential

Part B: open-label, cross-over

ELIGIBILITY:
Inclusion Criteria:

* Healthy, young, non-smoking men, weight ≥60 kg, and a body mass index (BMI) ≥18.5 kg/m2 and ≤30 kg/m2 at the Screening Visit.

Other in- and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (Safety and Tolerability) | From baseline to Day 9 (Part A and B)
  Based on the safety assessments (e.g. clinical safety laboratory tests, vital signs, weight and ECG parameters)

SECONDARY OUTCOMES:
AUC (0-inf) of Lu AG06479 | From pre-dose to Day 5 (Part A and B)
  Area under the Lu AG06479 concentration-time curve from time zero to infinity (AUC0-inf)
CL/F Lu AG06479 | From pre-dose to Day 5 (Part A and B)
  Oral clearance of Lu AG06479
Cmax Lu AG06479 | From pre-dose to Day 5 (Part A and B)
  Maximum observed plasma concentration for Lu AG06479

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance, Madison, Wisconsin, United States